CLINICAL TRIAL: NCT00300092
Title: Pediatric Fingertip Injuries: Do Prophylactic Antibiotics Alter Infection Rates?
Brief Title: Pediatric Fingertip Injuries:Are Antibiotics Required?
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Caroline Altergott, Assistant Professor of Pediatrics, Children's Hospital Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCI 99.156
Record Dates: First submitted 2006-03-06; First posted 2006-03-08 (Estimated); Last update posted 2015-04-20 (Estimated); Status verified 2015-04

CONDITIONS: Finger Injuries
MeSH Terms: conditions — Finger Injuries | interventions — Pharmaceutical Preparations; Cephalexin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No antibioitcs (No Intervention): Group 1 received no antibiotics
- Cephalexin (Active Comparator): Group 2 received cephalexin at 50 mg/kg divided 3 times daily for 7 days
  Interventions: Drug: Cepahlexin (drug)

INTERVENTIONS:
Drug: Cepahlexin (drug) — Cephalexin 50 mg/kg divided 3 times daily for 7 days
  Other Names: keflex
  Arms: Cephalexin

SUMMARY:
Study objective: Fingertip injuries are common in the pediatric population. Considerable controversy exists about whether prophylactic antibiotics are necessary after repair of such injuries. Our goals were to estimate the rate of bacterial infection among pediatric patients with distal fingertip injuries overall and to compare the rate of bacterial infections among subgroups treated with and without prophylactic antibiotics.

Methods: This was prospective randomized control study of pediatric patients presenting to an urban children's hospital with trauma to the distal fingertip requiring repair. Patients were randomized to two groups: those receiving prophylactic antibiotics (Cephalexin) and those who did not receive antibiotic therapy. Repairs were performed in a standardized fashion and all patients were re-evaluated in the same emergency department in 48 hours and by phone 7 days later. The primary outcome of this study was the incidence of infection.

DETAILED DESCRIPTION:
MATERIAL and METHODS Study design, Setting and Selection of Participants

This prospective randomized control trial was conducted at an urban children's hospital Emergency Department with 56,000 visits annually. The Institutional Review Board (IRB) approved the study prior to subject enrollment. The study period was from September 2000 to July 2004. All patients under 18 years of age presenting to the Emergency Department with a fingertip injury distal to the distal interphalangeal joint were eligible to participate. Patients were excluded from the study if the time from injury to repair was greater than eight hours, if the patients had diabetes, an oncologic disorder, an immune deficiency, a bleeding disorder, used steroids regularly, presented with a grossly contaminated wound, were currently taking antibiotics, or had a previous allergic reaction to cephalosporins.

The study was formulated as an equivalence trial to demonstrate non-inferiority of repair without versus with prophylactic antibiotics. The rate of infection 7 days after repair was the primary outcome variable. Determination of the target sample size was based on a combination of practicality and maximum difference between infection rates consistent with equivalence. It was judged feasible to enroll 160 subjects over the course of the study. Sample sizes of 80 per group would have 80% power to conclude with 95% certainty that the infection rates in the two groups were equivalent. This calculation is based on an upper 1-sided 95% confidence limit for the difference in infection rates, with percent infected of 6.25% in both groups, and the maximum allowable difference resulting in equivalence to be 10.6%.

Intervention

All wounds were treated following a standardized protocol.9, 10 First, the degree of injury was recorded. Fingertips were classified into one of five categories: no laceration (damage to nailbed), simple laceration, loss of skin or pulp, partial amputation or complete amputation. Subungal hematomas were drained by cautery. Hand x-rays were obtained to detect fractures, dislocations, or foreign bodies. Lacerations were irrigated with 500cc normal saline after a digital block with 1% lidocaine (no epinephrine). Devitalized tissue was removed. Skin lacerations and nail bed injuries were repaired with chromic gut. Xeroform gauze was then applied to the repaired finger and a bulky dressing secured. A tetanus booster was given if patient's immunizations were not up-to-date. At discharge study participants were given a standard wound care instruction sheet and a scheduled follow-up appointment at 48 hours. Subjects were told to return immediately to the same Emergency Department if they noticed signs or symptoms of infection, including the presence of redness, warmth, tenderness, swelling, discharge or fever.

All wounds were repaired by residents, fellows, and/or attending physicians in the Emergency Department. In-service training was provided in the Emergency Department prior to starting the study and periodically during the study period to assure consistency in the repair process. If the wound was repaired by a resident or fellow, the attending in the Emergency Department provided direct supervision.

After standard wound repair, eligible patients (and caregivers) were approached for enrollment. Interpreters were provided if the caregiver's or patient's primary language was not English. If caregivers and appropriate study subjects agreed, informed consent was obtained. Participants were then randomized to one of two groups using a randomization list prepared in advance with PROC PLAN within the Statistical Analysis System (SAS).11 Subjects assigned to Group 1 received no antibiotics after fingertip repair. Group 2 received prophylactic antibiotics (Cephalexin 50 mg/kg three times daily), upon discharge for 7 days. Cephalexin was chosen as the antibiotic of choice because the majority of wound infections are caused by gram positive organism (Staphylococcus and Streptococcus species). The full 7-day course of antibiotics was dispensed to study subjects prior to discharge. The cost of the antibiotics was covered by the General Clinical Research Center (GCRC).

A 48-hour follow-up visit was scheduled and the subject was told that one of the primary investigators would contact them by phone in 7 days. Subjects received instructions to keep their hand elevated, to keep the dressing clean and dry, to leave the dressings in place and to return to the Emergency Department immediately if signs or symptoms of wound infection developed.

At the follow-up visit and with the phone call, one of the three study investigators evaluated for the presence of infection, compliance with antibiotics, and wound healing. Infection was determined by the presence of erythema, tenderness, warmth, purulent discharge, regional lymphadenopathy, and fever. Subject compliance with the antibiotic regime was recorded at 48 hours and at 7 days after repair. Compliance was determined by phone follow-up asking the caregiver to measure the amount of antibiotic left in the bottle and asking for the number of doses administered.

Data Collection and Processing

Study data were collected at the initial visit by the physician repairing the wound. Data from the 48 hour and 7 day phone follow-up were collected by one of the three primary investigators. All data was recorded on a standardized data collection form and then entered into a computerized Microsoft Excel spreadsheet. All hospital charts were reviewed by the primary investigator at the close of the study for quality assurance purposes.

Statistical Methods

The two groups were compared for age, gender, time of injury, place of injury, mechanism of injury, finger involved, presence of fracture, complexity of injury, level of training of the treating physician, laceration experience of the treating physician, and number of sutures placed, using the 2-sample t-test or the Wilcoxon rank sum test for continuous variables and Fisher's exact test or a Chi squared test for categorical variables. The rate of infection 7 days after repair was calculated for each treatment group, along with exact binomial 95% confidence intervals. To assess the equivalence of the two treatments, the difference D = infection rate in the No Antibiotic Group minus infection rate in the Antibiotic Group was calculated. The upper limit of a 1-sided 95% confidence interval for D was used to estimate the maximum amount by which the infection rate without antibiotics may exceed that with prophylactic antibiotics. Additional analyses included comparison between dropouts and those who completed the study on demographic variables and wound and repair characteristics, and comparisons between those with and without infection to identify potential predictors of infection other than group assignment. NCSS 2004 software was used for equivalence testing.12 Statistical tests comparing group characteristics were 2-sided and considered significant for p<0.05, using the SAS software, version 8.11

DATA ANALYSIS

Characteristics of Study Subjects

A total of 146 subjects were initially enrolled in the study. The study was terminated earlier than expected because of staffing issues. Eleven participants were withdrawn prior to study completion. Those not completing the study included four subjects who could not be reached for phone follow-up, three subjects who received antibiotics during the study period for a reason other than infection of the fingertip, two subjects for whom insufficient data was available for analysis, one subject who received antibiotics prior to repair and one subject who requested to be withdrawn from the study prior to completion. These eleven subjects were significantly older than those who completed the study (6.0 +/- 3.8 vs. 3.1 +/- 2.7 years, p=0.001), but were similar on all other baseline characteristics. In addition, subjects were equally distributed between the 2 groups: 6/75 (8%) from Group 1(No Antibiotic) and 5/71 (7%) from Group 2(Antibiotic) (p=1.0).

A total of 135 subjects completed the study, 69 assigned to Group 1(No Antibiotic) and 66 assigned to Group 2(Antibiotic). Baseline characteristics of the two groups are shown in Table 1. Values tabulated are mean + s.d. for continuous variables and number and percent for categorical variables. No statistically significant differences on any baseline values were found between the two treatment groups. At the 7 day interview, the percent who reported consuming at least 75% of the prescribed doses was 86.2% (95% CI: 75.3%, 93.5%).

Results

At 7 days after repair, one subject in each treatment group had an infection. The subject in the No Antibiotic Group was treated with oral antibiotics and the subject in the Antibiotic Group was treated with intravenous antibiotics. Both made a full recovery. The infection rate (95% confidence interval) was 1.45% (0.04%, 7.81%) for the No Antibiotic Group and was 1.52% (0.04%, 8.16%) for the Antibiotic Group, not statistically significant (p=1.00). The upper limit of a 1-sided 95% confidence interval for the difference in rates was 4.9% indicating that there is a 5% chance that the infection rate in subjects not treated with antibiotics would exceed that of subjects treated with antibiotics by more than 4.9%.

Although the number of infections was too small for meaningful statistical comparisons, examination of the two infected cases revealed that the number of sutures was considerably larger than that among the uninfected subjects. The number of sutures for the two infected subjects was 8 and 9 (mean=8.5; standard deviation=0.7) and the mean (S.D.) for the uninfected subjects was 4.9 (2.0). After the completion of the study, chart review revealed four infections presenting beyond the seven-day window (Days 7-14), three in the Antibiotic Group and one in the No Antibiotic group. Interestingly, 41% of all wounds involved a fracture and none of these became infected.

ELIGIBILITY:
Inclusion Criteria:

* age 0-18 years
* fingertip injury distal to the distal interphalageal joint that requires repair

Exclusion Criteria:

* injury greater than 8 hours old
* diabetes
* oncologic disorder
* t-cell deficiency
* bleeding disorder
* chronic steriod use
* grossly contaminated wound
* allergy to Cephalexin
* current use of antibiotics

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 146 (Actual)
Dates: Start 2000-09; Primary Completion 2004-07 (Actual); Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
Pediatric Fingertip Injuries Do Prophylactic Antibiotics Alter Infection Rates | 4 years
  Incidence of infection in pediatric distal fingertip injuries that were treated with antibiotics and those that were not treated with antibiotics.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Altergott, MD, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Childrens Hospitla Los Angeles, Los Angeles, California, United States